CLINICAL TRIAL: NCT03439878
Title: The Acute Effects of Galactose Ingestion on Oral Fat Tolerance
Brief Title: Effect of Galactose Ingestion on Postprandial Lipemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Associate Professor, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MSES 16/17-011
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Cardiovascular Risk Factor; Lipemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Galactose; Glucose

STUDY DESIGN:
Intervention Model Description: Randomized, blinded crossover design.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and the researchers performing biochemical analyses will be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Galactose (Experimental): Ingestion of 0.75 g/kg body mass of d-galactose monohydrate co-ingested with cream to provide 1 g/kg body mass of fat.
  Interventions: Dietary Supplement: Galactose
- Glucose (Active Comparator): Ingestion of 0.75 g/kg body mass of dextrose monohydrate co-ingested with cream to provide 1 g/kg body mass of fat.
  Interventions: Dietary Supplement: Glucose

INTERVENTIONS:
Dietary Supplement: Galactose — Co-ingestion of d-galactose with a high-fat meal
  Arms: Galactose
Dietary Supplement: Glucose — Co-ingestion of d-glucose with a high-fat meal
  Arms: Glucose

SUMMARY:
This study aims to assess the postprandial triglyceride response to the ingestion of a high-fat meal with co-ingestion of either galactose, or glucose.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 to 35 years old
* Body mass index <30 kg/m2

Exclusion Criteria:

* Female
* Body mass index >29.9 kg/m2
* Any history of metabolic disease
* Allergies or intolerances to milk and/or cream

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Postprandial increase plasma triglyceride concentrations | 5 hours
  Incremental area under the curve (iAUC) of plasma triglyceride concentrations

SECONDARY OUTCOMES:
Postprandial plasma insulin concentrations | 5 hours
  Incremental area under the curve (iAUC) of plasma insulin concentrations
Postprandial plasma glucose concentrations | 5 hours
  Incremental area under the curve (iAUC) of plasma glucose concentrations
Postprandial plasma non-esterified fatty acid concentrations | 5 hours
  Postprandial area under the curve of non-esterified fatty acid concentrations
Postprandial plasma lactate concentrations | 5 hours
  Incremental area under the curve (iAUC) of plasma lactate concentrations
Postprandial subjective hunger ratings | 5 hours
  Postprandial area under the curve of hunger ratings measured by visual analogue scales (0-100 mm)
Postprandial subjective fullness ratings | 5 hours
  Postprandial area under the curve of fullness ratings measured by visual analogue scales (0-100 mm)
Postprandial subjective satisfaction ratings | 5 hours
  Postprandial area under the curve of satisfaction ratings measured by visual analogue scales (0-100 mm)
Postprandial prospective food consumption ratings | 5 hours
  Postprandial area under the curve of prospective food consumption ratings measured by visual analogue scales (0-100 mm)
Postprandial overall appetite ratings | 5 hours
  Postprandial area under the curve of overall appetite ratings measured by visual analogue scales (0-100 mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Raw data will be made available online upon publication in a peer-reviewed journal.

REFERENCES:
- [Derived] Watkins J, Simpson A, Betts JA, Thompson D, Holliday A, Deighton K, Gonzalez JT. Galactose Ingested with a High-Fat Beverage Increases Postprandial Lipemia Compared with Glucose but Not Fructose Ingestion in Healthy Men. J Nutr. 2020 Jul 1;150(7):1765-1772. doi: 10.1093/jn/nxaa105. PMID 32297937